CLINICAL TRIAL: NCT06228456
Title: Pharmacodynamic Effects of Low-dose Ticagrelor vs. Clopidogrel in Stable Patients Undergoing Elective Percutaneous Coronary Intervention Who Are At Risk of Peri-PCI Myocardial Infarction Using a Precision Medicine Tool
Brief Title: Effects of Low-dose Ticagrelor vs. Clopidogrel in Stable Patients Undergoing Elective Percutaneous Coronary Intervention
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Scott R. MacKenzie Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202302083
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease
Keywords: platelet reactivity; antiplatelet therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low-dose ticagrelor (Experimental): Stable CAD patients undergoing elective PCI treated with standard of care clopidogrel will be randomly assigned in a 1:1 fashion to either switch to ticagrelor or continue with clopidogrel.
  Interventions: Drug: Ticagrelor 60mg
- Clopidogrel (Active Comparator): Stable CAD patients undergoing elective PCI treated with standard of care clopidogrel will be randomly assigned in a 1:1 fashion to either switch to ticagrelor or continue with clopidogrel.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor 60mg — Patients in the ticagrelor arm will receive a 180 mg loading dose of ticagrelor followed by ticagrelor 60 mg bid maintenance dose for 30±5 days. Patients will maintain aspirin 81 mg once daily for the duration of the study.
  Other Names: Brilinta
  Arms: Low-dose ticagrelor
Drug: Clopidogrel — Patients in the clopidogrel arm will continue to receive clopidogrel 75 mg/daily for 30±5 days. Patients will maintain aspirin 81 mg once daily for the duration of the study.
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
The proposed study aims to assess the antiplatelet effects of more potent oral P2Y12 inhibition with low-dose ticagrelor (60 mg bid) compared with standard of care clopidogrel in patients with a high ABCD-GENE score (≥10). We hypothesize that ticagrelor is associated with better pharmacodynamic effects (i.e., lower platelet reactivity and high platelet reactivity rates) compared with clopidogrel in stable coronary artery disease patients undergoing percutaneous coronary intervention with a high ABCD-GENE score.

DETAILED DESCRIPTION:
Clopidogrel is the P2Y12 inhibitor of choice in patients with stable coronary artery disease (CAD) undergoing elective percutaneous coronary intervention (PCI). However, clopidogrel effects are subject to variability and 30-40% of patients have high platelet reactivity (HPR), which translates into higher rates of thrombotic complications. Despite the relative safety of PCI with new generation stents, peri-PCI thrombotic complications, including myocardial infarction and myocardial injury, are common in elective PCI. Importantly, these events are associated with poor prognosis, including cardiovascular mortality. The risk of peri-PCI myocardial infarction/myocardial injury has been in part attributed to HPR. A precision medicine tool integrating clinical (age, body mass index, chronic kidney disease and diabetes) and genetic (CYP2C19 loss-of-function allele status) factors called ABCD-GENE is able to identify HPR status. This score helps characterize patients at risk for peri-PCI thrombotic complications, who can thus potentially benefit from changes in antiplatelet treatment regimen. The new generation oral P2Y12 inhibitors prasugrel and ticagrelor are more potent than clopidogrel and associated with lower HPR rates and improved outcomes. Hence, these agents may be beneficial in reducing peri-PCI myocardial infarction/myocardial injury. Standard-dose ticagrelor (90 mg bid) provides more potent antiplatelet effect than clopidogrel in patients with ACS. Low-dose ticagrelor (60 mg bid) is beneficial in patients with prior myocardial infarction and has the potential of better bleeding profile compared to standard dose.This prospective randomized study aims to assess the antiplatelet effects of more potent oral P2Y12 inhibition with low-dose ticagrelor (60 mg bid) compared with standard of care clopidogrel in patients with a high ABCD-GENE score (≥10). We hypothesize that ticagrelor is associated with better PD effects (i.e., lower platelet reactivity and HPR rates) compared with clopidogrel in stable CAD patients undergoing PCI with a high ABCD-GENE score.

ELIGIBILITY:
Inclusion Criteria:

1. Stable CAD undergoing elective PCI;
2. Male or females, Age ≥ 18 years old;
3. Troponin negative before coronary angiography;
4. On treatment with low-dose aspirin (81mg od) and clopidogrel for at least 24 hours after index PCI;
5. ABCD-GENE score greater or equal than 10.

Troponin negative is defined as hs-cTn below the URL for the laboratory (Male < 22 ng/L; Female < 14 ng/L) or modestly positive hs-cTn (Male: 22-99 ng/L; Female: 14-99 ng/L) flat or decreasing from hour 0 to 3.

Exclusion Criteria:

1. Myocardial infarction at the time of index PCI;
2. On treatment with prasugrel or ticagrelor;
3. Documented hypersensitivity to clopidogrel;
4. Use of an intravenous antiplatelet therapy (i.e., cangrelor or GPI) in the prior 24 hours;
5. Concomitant therapy with strong CYP3A4 inhibitors or CYP3A4 substrates;
6. Use of oral anticoagulant therapy;
7. History of previous intracerebral bleed at any time;
8. Active pathological bleeding;
9. Documented hypersensitivity to ticagrelor;
10. Increased risk of bradycardic events (e.g., known sick sinus syndrome, second or third degree AV block or previous documented syncope suspected to be due to bradycardia) unless treated with a pacemaker;
11. Known severe liver disease;
12. Known platelet count <80x106/mL;
13. Known hemoglobin <9 g/dL;
14. Women of child-bearing potential (i.e., those who are not chemically or surgically sterilized or who are not post-menopause) who are not willing to use a medically accepted method of contraception that is considered reliable in the judgment of the investigator OR who have a positive pregnancy test at enrollment or randomization OR women who are breast-feeding.
15. Inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
P2Y12 reaction units (PRU) | 30 days
  The primary endpoint will be platelet reactivity measured by VerifyNow PRU

SECONDARY OUTCOMES:
Maximum platelet aggregation | 30 days
  Platelet aggregation will be measured using light transmittance aggregometry (LTA) with 20 μmol/L ADP as stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Franchi, MD, Principal Investigator — Univesrsity of Florida
Locations (1):
- University of Florida Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No